CLINICAL TRIAL: NCT00082394
Title: A Phase IV Randomized, Multicenter, Open-Label Study to Compare the Safety, Tolerability and Efficacy of Trizivir (Abacavir 300mg, Lamivudine 150mg, and Zidovudine 300mg) BID vs Combivir (Lamivudine 150mg and Zidovudine 300mg) BID Plus Atazanavir 400mg QD in Antiretroviral Naive HIV-1 Infected Subjects Over 48 Weeks
Brief Title: A Study Comparing The Safety, Tolerability and Efficacy of Trizivir VS Combivir & Atazanavir In Subjects With HIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 100327
Record Dates: First submitted 2004-05-06; First posted 2004-05-10 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Infection, Human Immunodeficiency Virus I; HIV Infection
Keywords: safety; drug efficacy; TRIZIVIR; tolerability; COMBIVIR; HIV; atazanavir
MeSH Terms: conditions — Infections; HIV Infections | interventions — abacavir, lamivudine, and zidovudine drug combination; Atazanavir Sulfate; lamivudine, zidovudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Trizivir
Drug: atazanavir
Drug: Combivir
  Other Names: atazanavir; Trizivir

SUMMARY:
The aim of this study was to assess whether TRIZIVIR, administered twice-daily was as safe, tolerable and efficacious as a combination of the drugs COMBIVIR administered twice-daily and atazanavir administered once daily. Over the course of 48 weeks, various parameters that measure safety, tolerability and efficacy of the investigational drugs were measured and compared.

DETAILED DESCRIPTION:
A Phase IV Randomized, Multicenter, Open-Label Study to Compare the Safety, Tolerability and Efficacy of Trizivir (abacavir 300mg, lamivudine 150mg, and zidovudine 300mg) BID vs Combivir (lamivudine 150mg and zidovudine 300mg) BID plus atazanavir 400mg QD in Antiretroviral Naive HIV-1 Infected Subjects over 48 Weeks

ELIGIBILITY:
Inclusion criteria:

* Adults with documented HIV-1 infection.
* Past use of HIV drugs must have been less than 15 days.
* Plasma HIV-1 RNA between 500 and 20,000 copies/mL.
* CD4+ cell count greater than 100 cells/mm3.
* Willing/able to provide written informed consent.

Exclusion criteria:

* Have AIDS at screening.
* Pregnant or breastfeeding.
* Underlying medical conditions considered to be significant for this protocol.
* Participating in other investigational drug trials.
* In the opinion of the investigator, would be unable to complete 48 weeks of dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-04-26 (Actual); Primary Completion 2006-03-01 (Actual); Study Completion 2006-03-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was drug efficacy, measured as the proportion of study subjects who had plasma HIV-1 RNA less than 50 copies/mL at week 48 and did not meet the definition of virologic failure through this timepoint. | 48 Weeks

SECONDARY OUTCOMES:
% patients with plasma HIV-1 RNA <50 and <400 copies/mL at weeks 24 & 48; Change from BL in plasma HIV-1 RNA and CD4+ measures; AEs; Time to virologic failure | 48 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (40):
- United States (38):
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Beach, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, East Orange, New Jersey
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Voorhees Township, New Jersey
  - GSK Investigational Site, Mount Vernon, New York
  - GSK Investigational Site, Valhalla, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, West Reading, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Harlingen, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Hampton, Virginia
- Mexico (2):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León

REFERENCES:
- [Derived] Kumar PN, Salvato P, LaMarca A, DeJesus E, Patel P, McClernon D, Florance A, Shaefer MS. A randomized, controlled trial of initial anti-retroviral therapy with abacavir/lamivudine/zidovudine twice-daily compared to atazanavir once-daily with lamivudine/zidovudine twice-daily in HIV-infected patients over 48 weeks (ESS100327, the ACTION Study). AIDS Res Ther. 2009 Apr 9;6:3. doi: 10.1186/1742-6405-6-3. PMID 19358725